CLINICAL TRIAL: NCT05939557
Title: Effects of Kinesio Taping vs Jones Technique on Myofascial Trigger Points in Cervicalgia: a Pilot Study of a Randomised Control Trial.
Brief Title: Effects of Kinesio Taping vs Jones Technique on Myofascial Trigger Points in Cervicalgia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Blanca González Sanchez (Other)
Responsible Party: Sponsor-Investigator, Blanca González Sanchez, PHD, University of Extremadura
Organization: University of Extremadura (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 01/2015
Record Dates: First submitted 2023-06-10; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-06

CONDITIONS: Cervicalgia
Keywords: Cervicalgia; cinta de kinesio; Técnica de Jones; fisioterapia; puntos de activación.
MeSH Terms: conditions — Neck Pain | interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Jones technique group (Experimental): Performs Jones technique 12 participants.
  Interventions: Procedure: Jones technique
- kinesio tapping group (Experimental): Performs kinesiotape 14 participants.
  Interventions: Device: Kinesiotape
- combined therapy group (Experimental): Performs Jones technique and kinesiotape 12 participants.
  Interventions: Procedure: Jones technique; Device: Kinesiotape

INTERVENTIONS:
Procedure: Jones technique — is a gentle soft tissue manipulation consisting of a passive procedure that positions the body in a position of comfort to release tissue that compresses or shortens the body structure (muscle contraction and joint dysfunction)
  Arms: Jones technique group; combined therapy group
Device: Kinesiotape — KT has an S-shaped glue, which lifts the skin, thus improving blood and lymphatic circulation, with the intention of relieving pain and improving musculoskeletal diseases especially in sports
  Arms: combined therapy group; kinesio tapping group

SUMMARY:
A large number of workers in different sectors suffer from musculoskeletal neck disorders, which are the most common work-related illness in Europe. A multitude of combinations of techniques can be used to treat these conditions, including recorded film and the Jones technique. This pilot study examines the efficacy of Kinesio taping and the Jones technique in improving pain, joint range of motion and muscle tension in active subjects with latent myofascial trigger points. A clinical trial was conducted with 38 patients with neck pain. The sample was randomly distributed into three groups: a Jones technique group, a kinesio taping group and a combined therapy group in which both techniques were performed. The duration of treatment was 4 weeks, with a follow-up of 2 weeks. Cervical spine joint range of motion, pain and functional disability were assessed with the goniometer, the visual analogue scale, the pressure algometer and the cervical disability index.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of latent PGM in the upper trapezius
* Have been working for more than 6 months in the center or company
* Work more than 4 hours a day with the computer
* Be over 18 years of age and under 64 years of age

Exclusion Criteria:

* Diagnosis of fibromyalgia
* Having suffered a cervical sprain
* Diagnosis of radiculopathy, cervical spine surgery
* Medical contraindications to neuromuscular bandaging or Jones technique
* Diseases such as diabetes and cancer, pregnancy, and any other pathology that produces neck pain other than that specified in the objective of the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2015-04-01 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline VAS at 4 weeks of treatment and at the 2-week follow-up | time 0, after 4 weeks of treatment, and at the 2-week follow-up
  Visual Analogue Scale (VAS), consisting of a 10 cm line representing the continuous spectrum of painful experience. Only at the ends appear descriptions, "no pain" at one end and "worst pain imaginable" at the other, with no other description along the line. The subject will subjectively estimate his or her level of pain by indicating it on the ruler
Change from Baseline UDP at 4 weeks of treatment and at the 2-week follow-up | time 0, after 4 weeks of treatment, and at the 2-week follow-up
  Measurement of the pressure pain threshold (UDP) This is performed using a pressure algometer that aims to objectify the ability of muscle fibers to adapt to compression on underlying planes
Change from Baseline NDI at 4 weeks of treatment and at the 2-week follow-up | time 0, after 4 weeks of treatment, and at the 2-week follow-up
  Neck Disability Index (NDI), a questionnaire for self-assessment of function and activity disability in patients with neck pain. It consists of 10 items referring to functional activities, pain intensity, concentration and headache. The maximum score is 50 points, so that the higher the score the worse the function
Change from Baseline GONIOMETER at 4 weeks of treatment and at the 2-week follow-up | time 0, after 4 weeks of treatment, and at the 2-week follow-up
  Goniometer, instrument used for the study of joint mobility (MA). Cervical flexion, right and left lateralizations, and right and left rotations were evaluated. Each measurement was made three times with a separation of 30 seconds in time, taking the average between the three measurements.

IPD SHARING:
Plan to Share IPD: No